CLINICAL TRIAL: NCT04357418
Title: Psychological Outcome of COVID-19 Lockdown on Psychiatric Hospital Staff and Close Relatives (ICOS)
Brief Title: Psychological Outcome of COVID-19 Lockdown on Psychiatric Hospital Staff and Close Relatives
Acronym: ICOS
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Clémence ISAAC, Psychologist, Centre hospitalier de Ville-Evrard, France
Other Study IDs: 10477M-ICOS
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Anxiety State; COVID-19; Isolation, Social; Health Personnel Attitude
Keywords: anxiety; depression; anger; quarantine; health care workers
MeSH Terms: conditions — Anxiety Disorders; COVID-19; Social Isolation; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hospital staff
  Interventions: Other: it is a survey
- close relatives.
  Interventions: Other: it is a survey

INTERVENTIONS:
Other: it is a survey — this interview can be carried out face to face or remotely.

SUMMARY:
The purpose of the investigators is to study the psychological impact of the COVID-19 lockdown on the members of the Ville Evrard Hospital staff and their close relatives, and to identify potential lockdown conditions that could increase anxiety, anger and depressive symptoms in this population.

ELIGIBILITY:
Inclusion Criteria:

* For hospital staff: Adult members of the Ville Evrard Hospital staff (trainees or employees) willing to participate to at least one survey during the COVID lockdown.
* For close relatives: Adult relatives of the Ville Evrard Hospital staff members, living or not with them.

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is about hospital staff and close relatives
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
State Anxiety assessed by the State-Trait Anxiety Inventory (STAI) | Up to one month and a half after the beginning of the lockdown (From March 17th to May 1st 2020)
  The "State Trait Inventory Anxiety" is widely used both in practice and in clinical research. It consists of separate scales for assessing state (STAI form Y-A) and trait (STAI form Y-B). Each of the scales includes 20 items, the E scale to assess how subjects feel at the time, the T scale to capture how subjects feel generally.The STAI is intended for self-administration. It can be completed individually or in a group.
State Anxiety assessed by the State-Trait Anxiety Inventory (STAI) | Up to one month and a half after the end of the lockdown (from May 11th to June 25th)
  The "State Trait Inventory Anxiety" is widely used both in practice and in clinical research. It consists of separate scales for assessing state (STAI form Y-A) and trait (STAI form Y-B). Each of the scales includes 20 items, the E scale to assess how subjects feel at the time, the T scale to capture how subjects feel generally.The STAI is intended for self-administration. It can be completed individually or in a group.

SECONDARY OUTCOMES:
Visual numeric scales assessing anger and stress the ongoing week. | Up to one month and a half after the beginning of the lockdown (From March 17th to May 1st 2020)
  1 to 7 Likert scales. Anger scale going from "No anger, at no time" to "strong and sustained anger". Stress scale going from "No stress, at no time" to "strong and sustained stress".
Visual numeric scales assessing anger and stress the ongoing week. | Up to one month and a half after the end of the lockdown (from May 11th to June 25th)
  1 to 7 Likert scales. Anger scale going from "No anger, at no time" to "strong and sustained anger". Stress scale going from "No stress, at no time" to "strong and sustained stress".
Beck Depression Inventory | Up to one month and a half after the beginning of the lockdown (From March 17th to May 1st 2020)
  The tool provides a quantitative estimate of the intensity of depressive feelings.
Beck Depression Inventory | Up to one month and a half after the end of the lockdown (from May 11th to June 25th)
  The tool provides a quantitative estimate of the intensity of depressive feelings.

CONTACTS AND LOCATIONS:
Overall Officials: Clemence ISAAC, PhD, Principal Investigator — CH Ville Evrard; Dominique JANUEL, Pr, Study Director — CH Ville Evrard
Locations (1):
- URC Ville Evrard, Neuilly-sur-Marne, France

IPD SHARING:
Plan to Share IPD: Undecided